CLINICAL TRIAL: NCT06495307
Title: A PHASE I PROSPECTIVE OPEN LABEL STUDY ASSESSING THE SAFETY & EFFICACY OF RHPRG4 (450 µG/ML RECOMBINANT HUMAN PROTEOGLYCAN 4) FOR THE TREATMENT OF OCULAR GRAFT-VERSUS-HOST DISEASE (OGVHD)
Brief Title: RHPRG4 FOR THE TREATMENT OF OCULAR GRAFT-VERSUS-HOST DISEASE (OGVHD)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Efficacy signal substantial enough to more to larger study
Sponsor: Lubris Bio Pty Ltd (Industry)
Collaborators: Lubris, LLC (Unknown); Sydney Eye Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RHPRG4-OGVHD-001
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Ocular Graft-versus-host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: rhPRG4

INTERVENTIONS:
Drug: rhPRG4 — Sterile isotonic aqueous solution containing rhPRG4 (450 µg/mL) for topical administration, 10 mM sodium phosphate, 150 mM sodium chloride & 0.01% polysorbate 20 at pH 7.2. In all subjects, both eyes will be treated

SUMMARY:
rhPRG4-GVHD-001 is a prospective multi-center study conducted in Australia to evaluate the safety and efficacy of topically-applied rhPRG4 in subjects with moderate to severe dry eye secondary to chronic GVHD.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis and Main Criteria for Inclusion:

All to be queried and checked at the screening visit (V1):

1. Subjects 18 years of age or older;
2. Subjects diagnosed with oGVHD for at least 3 months (current use of artificial tears for the treatment of GVHD);
3. VAS Eye Dryness (100-point scale) score ≥ 60 mm;
4. Tear Osmolarity ≥ 312 in either eye;
5. Corneal staining score with fluorescein ≥ 2 using the Oxford scale in the worst performing eye; staining must include quadrants beyond only inferior or superior staining;
6. Only subjects who satisfy all Informed Consent requirements may be included in the study.

Exclusion Criteria:

Diagnosis and Main Criteria for Exclusion:

1. Evidence of an active ocular infection in either eye;
2. History or presence of ocular surface disorders not related to oGVHD in either eye, including but not limited to significant conjunctivochalasis, superior limbic keratoconjunctivitis, limbal stem cell deficiency, allergic conjunctivitis, giant papillary conjunctivitis, atopic keratoconjunctivitis, anterior basement membrane dystrophies, neurotrophic keratitis, corneal dystrophy, exposure keratitis and moderate to severe blepharitis;
3. History of any ocular surgery (including laser or refractive surgical procedures) in either eye within 90 days before study enrollment. Ocular surgery will not be allowed during the study treatment period and elective ocular surgery procedures should not be planned during the duration of the follow-up period;
4. Initiation of new therapeutic modalities within 30 days of recruitment;
5. Artificial rescue tears are allowed as long as they are recorded in a diary;
6. Known hypersensitivity to one of the components of the study or procedural medications;
7. Participation in another clinical study at the same time as the present study or within 60 days of screening/baseline visit;
8. History of drug, medication or alcohol abuse or addiction;
9. Females of childbearing potential (those who are not surgically sterilized or post-menopausal for at least 1 year) are excluded from participation in the study if they meet any one of the following conditions:

   1. are currently pregnant or,
   2. have a positive result on the urine pregnancy test at the Screening/Baseline Visit or,
   3. intend to become pregnant during the entire course of and 30 days after the study treatment periods, or,
   4. are breast-feeding or,
   5. not willing to use highly effective birth control measures, such as: Hormonal contraceptives - oral, implanted, transdermal, or injected and/or mechanical barrier methods, during the entire course of and 30 days after the study treatment periods.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2025-02-14 (Actual); Primary Completion 2025-03-22 (Actual); Study Completion 2025-03-22 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of rhPRG4 using the average VAS score assessing subjects' eye dryness (Question: Rate the dryness of your eye; anchors: 0 = no discomfort, 100 = maximal discomfort) at Day 28 | 28
To assess the efficacy of rhPRG4 using the total corneal staining with fluorescein (Oxford Scale) at Day 28 | 28
To assess the safety of rhPRG4 by observation of the frequency and severity of treatment-emergent adverse events | 28

SECONDARY OUTCOMES:
To assess the efficacy of rhPRG4 using the average VAS score for foreign body sensation, burning/stinging, itching, pain, sticky feeling, blurred vision and photophobia and total VAS (anchors: not at all & very) | 28
To assess the efficacy of rhPRG4 using the maximum inter-eye tear osmolarity: max(OU) | 28
To assess the efficacy of rhPRG4 using the absolute difference in inter-eye tear film breakup time (TBUT): min(OU)osmolarity: abs(OD - OS) | 28
To assess the efficacy of rhPRG4 using the number of instillations of rescue artificial tear per day | 28
To assess the efficacy of rhPRG4 using a patient questionnaire | 28
To assess the efficacy of rhPRG4 by NIH Eye Score | 28
To assess the safety of rhPRG4 by observation of the Best Corrected Visual Acuity (BCVA) | 28
To assess the safety of rhPRG4 by observation of signs evaluated by slit lamp (SLE) | 28
To assess the safety of rhPRG4 by observation of intraocular pressure (IOP) | 28

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Sydney Eye Hospital, Sydney, New South Wales
  - OTA, Brisbane, Queensland

IPD SHARING:
Plan to Share IPD: No